CLINICAL TRIAL: NCT02802293
Title: Treatment of Depression With Connectivity Guided Robotically Delivered Repetitive Transcranial Magnetic Stimulation
Brief Title: Treatment of Depression With Connectivity Guided Robotically Delivered rTMS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study temporarily suspended due to COVID-19 pandemic then closed due to low enrollment numbers
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: IKARE Mood, Trauma, Recovery Clinic (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HSC20160129H; HSC20160129H (Other: UTHSCSA)
Record Dates: First submitted 2016-06-13; First posted 2016-06-16 (Estimated); Results first posted 2022-08-25 (Actual); Last update posted 2022-08-25 (Actual); Status verified 2022-06

CONDITIONS: Major Depressive Disorder
Keywords: Repetitive Transcranial Magnetic Stimulation; Major Depressive Disorder
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Transcranial Magnetic Stimulation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (3):
- Standard rTMS Aiming (Active Comparator): Active repetitive transcranial magnetic stimulation (rTMS) will be delivered to the left DLPFC using the standard aiming strategy with the rTMS coil positioned using a robotic arm. In this arm, rTMS will be delivered at 10 Hz in 4 sec trains with 26 sec inter-train intervals, 37.5 minutes/session (i.e. 3,000 pulses/session), 5 sessions/week, for 4 weeks.
  Interventions: Device: repetitive transcranial magnetic stimulation; Device: robotic arm
- Anterior DLPFC targeting (Active Comparator): Active rTMS will be delivered to the left anterior DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm. In this arm, rTMS will be delivered at 10 Hz in 4 sec trains with 26 sec inter-train intervals, 37.5 minutes/session (i.e. 3,000 pulses/session), 5 sessions/week, for 4 weeks.
  Interventions: Device: repetitive transcranial magnetic stimulation; Device: robotic arm
- Posterior DLPFC targeting (Active Comparator): Active rTMS will be delivered to the left posterior DLPFC using connectivity-based, image-guided aiming with the rTMS coil positioned using a robotic arm. In this arm, rTMS will be delivered at 10 Hz in 4 sec trains with 26 sec inter-train intervals, 37.5 minutes/session (i.e. 3,000 pulses/session), 5 sessions/week, for 4 weeks.
  Interventions: Device: repetitive transcranial magnetic stimulation; Device: robotic arm

INTERVENTIONS:
Device: repetitive transcranial magnetic stimulation — The MagPro R30 is an advanced, high performance magnetic stimulator designed primarily for non-invasive clinical use. The non-invasive brain stimulation system will be used to deliver repetitive electromagnetic pulses in this research study's treatment of major depressive disorder.
  Other Names: rTMS
Device: robotic arm — This robotic system is based on a commercially available neurosurgical robot. The robot is mounted on a mobile (i.e. retractable wheels) cart which holds the robot controller and the TMS power supply and pulse-generation computer. The robotic system will be used for TMS coil positioning/targeting.

SUMMARY:
The purpose of this study is to determine the clinical effects (if any) of connectivity-guided repetitive transcranial magnetic stimulation (rTMS) in the treatment of major depressive disorder (MDD) to provide clues about the ideal neural networks to target for more robust clinical outcomes, and to identify potential biomarkers of treatment response including changes in brain network connectivity.

DETAILED DESCRIPTION:
The investigators propose a randomized, double-blind, 4-week trial of TMS to the left dorsolateral prefrontal cortex (DLPFC) for subjects with MDD all of whom at the patient's treatment clinic are concurrently receiving pharmaceutical and psychotherapeutic interventions. Arm 1 delivers active rTMS to the left DLPFC using the standard aiming strategy. Arm 2 delivers active rTMS to the left anterior DLPFC using connectivity-based, image-guided aiming. Arm 3 delivers active rTMS to the left posterior DLPFC using connectivity-based, image-guided aiming. In all three arms, rTMS is administered in an image-guided, robotically-positioned TMS (irTMS) manner to ensure therapist blinding and equivalent subject experiences across arms. In all three arms, the following stimulation protocol will be used: 10 Hz irTMS delivered in 4 sec trains with 26 sec inter-train intervals, 37.5 minutes/session (i.e. 3,000 pulses/session), 5 sessions/week, for 4 weeks. Neuroimaging will be used both for treatment planning and to characterize any TMS-induced network plasticity using resting-state functional magnetic resonance imaging (rs-fMRI) at week 4 of each treatment arm. Clinical assessments will be administered weekly throughout treatment (weeks 1-4) at the patient's treatment clinic. Additional psychological tests will be performed at UT Health-San Antonio's Research Imaging Institute (RII) at the baseline and post-treatment visits in order to track patient progress.

ELIGIBILITY:
Inclusion Criteria:

1. Males or females with MDD receiving treatment at the iKare Mood Trauma Recovery Clinic between the ages of 18-65 years;
2. Meeting the fifth edition of the Diagnostic and Statistical Manual of Mental Disorders (DSM-V) criteria for MDD as determined using the Mini-International Psychiatric Interview (MINI)
3. Meeting the Patient Health Questionnaire-9 (PHQ-9 > 14) and/or the Structured Interview Guide for the Montgomery-Ashberg Depression Rating Scale (SIGMA>18) criteria for treatment resistance in MDD despite completing at least one adequate trial of an Selective Serotonin Reuptake Inhibitor (SSRI) or Serotonin-Norepinephrine Reuptake Inhibitor (SNRI) at an FDA-recommended dose for at least 6-8 weeks.
4. Subjects on SSRIs or other antidepressants, hypnotic medications including modulators of Gamma-Aminobutryic Acid (GABA)-A receptor function, trazodone, atypical neuroleptic or other psychotropic medications such as prazosin may enter the study if they are deemed to be on a stable dose of their medication.
5. Able to provide written informed consent.
6. Able to read and write English.

Exclusion Criteria:

1. Subjects with a diagnostic history of bipolar disorder, schizophrenia or schizoaffective disorder or currently exhibiting psychotic features as confirmed by MINI.
2. Serious, active suicidal risk as assessed by evaluating psychiatrist. Serious active suicidal risk is determine as imminent risk of suicide reflected in a subject having a plan and intent to end his or her life. History of suicidality in itself is not exclusion for participation in this protocol so long as the evaluating psychiatrist determines that there is an absence of serious active suicidal risk and the means to keep subjects safe.
3. Substance use disorder during the 3 months prior to screening; except for Mild or Moderate Alcohol Use Disorder according to DSM-V criteria.
4. Any history or signs of serious medical or neurological illness including seizure disorders. Except for seizures, a subject with a clinical abnormality may be included only if the study clinician considers the illness will not introduce additional risk and will not interfere with the study procedures.
5. Females will be excluded if they are pregnant (i.e. positive pregnancy test identified after their intake at the treatment clinic).
6. History of traumatic brain injury (TBI) with loss of consciousness for 20 minutes or more as determined by the Brief Traumatic Brain Injury Screen (TBI Screening Tool).
7. Any history or signs of metal objects (e.g. surgical clips, cardiac pacemakers, metal implants, etc.) in the body at the time of screening. MRI can have risks for persons with foreign bodies implanted in their body.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-08-17 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-03-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Felipe S Salinas, Ph.D., Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- Ikare, Mood, Trauma, Recovery Clinic, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: No
There is no plan to share individual participant data at this time.

REFERENCES:
- [Background] O'Reardon JP, Solvason HB, Janicak PG, Sampson S, Isenberg KE, Nahas Z, McDonald WM, Avery D, Fitzgerald PB, Loo C, Demitrack MA, George MS, Sackeim HA. Efficacy and safety of transcranial magnetic stimulation in the acute treatment of major depression: a multisite randomized controlled trial. Biol Psychiatry. 2007 Dec 1;62(11):1208-16. doi: 10.1016/j.biopsych.2007.01.018. Epub 2007 Jun 14. PMID 17573044

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Started | 1 | 2 | 3
Completed | 0 | 1 | 1
Not Completed | 1 | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting | Total
Number analyzed (Participants) | 1 | 2 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 1 | 2 | 2 | 5
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 3 | 4
  Male | 1 | 1 | 0 | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1 | 2
  Not Hispanic or Latino | 1 | 1 | 2 | 4
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 2 | 3 | 6

OUTCOME MEASURES:

1. Primary Outcome: Change in Depression Severity (MADRS)
Description: Measured by the Montgomery-Ashberg Depression Rating Scale. This is a 10-item diagnostic questionnaire with an overall score range from 0 to 60. A higher score indicates more severe depression:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
Time Frame: Baseline to four weeks (the conclusion of rTMS treatment)
Population: Discrepancies in the number of participants analyzed for this outcome measure occur because of patient withdrawals from treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Number analyzed (Participants) | 0 | 1 | 1
units on a scale
  baseline |  | 32 (0) | 43 (0)
  4 weeks |  | 2 (0) | 46 (0)

2. Secondary Outcome: Change in Depression Severity (MADRS)
Description: as for outcome 1
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: Discrepancies in the number of participants analyzed for this outcome measure occur because patients did not respond to follow-up calls.
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Clinically Significant Response (MADRS)
Description: Defined as greater than or equal to a 50% decrease in the Montgomery-Ashberg Depression Rating Scale. This is a 10-item diagnostic questionnaire with an overall score range from 0 to 60. A higher score indicates more severe depression:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
Time Frame: Baseline to four weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Number analyzed (Participants) | 0 | 1 | 1
Participants |  | 1 | 0

4. Secondary Outcome: Clinically Significant Response (MADRS)
Description: as for outcome 3
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 2
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Number analyzed (Participants) | 0 | 0 | 0

5. Secondary Outcome: Remission From Depression (MADRS)
Description: Defined as Montgomery-Ashberg Depression Rating Scale score less than or equal to 10. This is a 10-item diagnostic questionnaire with an overall score range from 0 to 60. A higher score indicates more severe depression:
  0 to 6 - normal/symptom absent 7 to 19 - mild depression 20 to 34 - moderate depression >34 - severe depression.
Time Frame: Baseline to four weeks (the conclusion of rTMS treatment)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Number analyzed (Participants) | 0 | 1 | 1
Participants |  | 1 | 0

6. Secondary Outcome: Remission From Depression (MADRS)
Description: as for outcome 5
Time Frame: Baseline to sixteen weeks (twelve weeks after the conclusion of rTMS treatment)
Population: as for outcome 2
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Functional Connectivity Changes of the Targeted Brain Network(s) Following rTMS Treatment
Description: resting-state fMRI scan will also be used to assess, network-specific functional connectivity differences between each subject's pre-treatment and post-treatment scans.
  The purpose of the Z score is to "standardize" distributions so that each has a mean of 0, and standard deviation as 1, so we can then make comparisons.
  Standard Score, the "Z-Score": A way to make a comparison between values on two different normal curves by converting the values to the number of standard deviations above or below the mean.
Time Frame: Baseline to four weeks (the conclusion of rTMS treatment)
Population: Functional brain connectivity to the sub-genual cingulate (SGC) cortex compared between the groups (in participants with 20 treatment sessions) at baseline and 4 weeks.
Measure: Number; unit: z-score
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
Number analyzed (Participants) | 0 | 1 | 1
z-score |  | -2.35 | 1.86

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Standard rTMS Aiming | Anterior DLPFC Targeting | Posterior DLPFC Targeting
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/2 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/2 | 0/3
Other Adverse Events (participants affected / at risk) | 1/1 | 1/2 | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Standard rTMS Aiming (N=1) | Anterior DLPFC Targeting (N=2) | Posterior DLPFC Targeting (N=3)
Headache (General disorders) | 1 (4) | 1 (15) | 1 (8)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/93/NCT02802293/Prot_SAP_002.pdf